CLINICAL TRIAL: NCT03865680
Title: Effect of Casein Phosphopeptide Amorphous Calcium Phosphate Fluoride Varnish on Remineralization of White Spot Lesion in Primary Teeth (Randomized Clinical Trial)
Brief Title: Effect of Casein Phosphopeptide Amorphous Calcium Phosphate Fluoride Varnish on Remineralization of White Spot Lesion in Primary Teeth
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nourhan M.Aly (Other)
Collaborators: Alexandria University (Other)
Responsible Party: Sponsor-Investigator, Nourhan M.Aly, Clinical Instructor and statistician, University of Alexandria
Organization: University of Alexandria (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CPP-ACP FV on remineralization
Record Dates: First submitted 2019-03-04; First posted 2019-03-07 (Actual); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: White Spot Lesion
Keywords: Fluoride varnish; Casein; MI varnish
MeSH Terms: interventions — casein phosphopeptide-amorphous calcium phosphate nanocomplex; sodium fluoride topical preparation; Bifluorid 12

STUDY DESIGN:
Intervention Model Description: The study is a double blind randomized controlled clinical trial, with a 1:1 allocation ratio. Subjects are randomly assigned using a computer -generated list of random numbers to one of the two arms (MI varnish, Duraphat fluoride varnish).
Who Masked: Participant, Outcomes Assessor
Masking Description: The Participants and the statistician are blinded to the treatment groups. The operator will not be blinded to the treatment as the test group will receive MI varnish while the control group will receive Duraphat varnish.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MI varnish (Experimental): MI Fluoride varnish: 5% sodium fluoride varnish water based, sugar free containing RecaldentTM (CPP-ACP) (GC AMERICA INC.3737 West 127th Street, Alsip, IL 60803 U.S.A). The varnish will be applied at baseline 2 and 4 weeks on the whole set of teeth of the participants with partial cotton roll isolation , saliva ejector and according to the manufacturer's instructions. Participants will receive oral hygiene instructions, prophylaxis without paste.
  Interventions: Drug: CPP-ACP
- Duraphat Fluoride varnish (Active Comparator): Duraphat Fluoride: varnish 5% sodium fluoride varnish (Colgate, New York, N.Y.). The varnish will be applied at baseline 2 and 4 weeks on the whole set of teeth of the participants with partial cotton roll isolation , saliva ejector and according to the manufacturer's instructions. Participants will receive oral hygiene instructions, prophylaxis without paste.
  Interventions: Drug: Duraphat

INTERVENTIONS:
Drug: CPP-ACP — The fluoride varnish applications will be applied with identical intensive protocols every 2 weeks for 6 weeks. The application of will be according to manufacturer's instructions.
  Other Names: MI varnish; Casein phosphopeptide-amorphous calcium phosphate fluoride varnish
  Arms: MI varnish
Drug: Duraphat — The fluoride varnish applications will be applied with identical intensive protocols every 2 weeks for 6 weeks. The application of will be according to manufacturer's instructions.
  Other Names: Sodium Fluoride varnish
  Arms: Duraphat Fluoride varnish

SUMMARY:
The aim of this study is to evaluate the effectiveness of Casein phosphopeptide-amorphous calcium phosphate fluoride varnish (CPP-ACP FV) in comparison to fluoride varnish (FV) as a remineralizing agent for white spot lesions in primary teeth (WSLs).

DETAILED DESCRIPTION:
The study is a two parallel arms double blinded randomized controlled clinical trial. A total of 180 WSL in primary teeth in chikdren aged 2-5 y and satisfying the inclusion criteria were selected. Patients will be randomly allocated into 2 groups allocated to two varnishes: study group: CPP-ACP FV (MI varnish), Control group FV (Duraphat). Both fluoride varnishes applications are applied with identical intensive protocols every 2 weeks for 6 weeks. The application of each varnish will be according to manufacturer's instructions. The operator is not blinded to treatment type. Only the participants and statistician are blinded to treatment groups. The whole sample (N=180) will be followed up at 6 weeks and at 18 and 30 weeks for Visio-tactile assessment and DIAGNOdent measurements

ELIGIBILITY:
Inclusion Criteria:

* Healthy children with no systemic diseases.
* High caries risk children with the presence of at least one visible active WSL in primary teeth with ICDAS II score of 1,2 or 3
* Completion of a parental consent to participate in the study.

Exclusion Criteria:

* Selected tooth with cavitated lesion.
* Selected tooth with enamel defects.
* Participants allergic to milk products.

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 180 (Actual)
Dates: Start 2019-04-28 (Actual); Primary Completion 2020-03-25 (Actual); Study Completion 2020-04-10 (Actual)

PRIMARY OUTCOMES:
Oral hygiene index (OHI-S) assessment | Baseline
  For primary dentition, the modified version of the OHI-S by Miglani et al will be used, it is divided into two scores debris index and calculus index only the debris index will be used in which the index teeth are: The buccal surface of maxillary right second molar (tooth 55), The buccal surface of the maxillary right central incisor (tooth 51), The buccal surface maxillary left second molar (tooth 65), The lingual surface of the mandibular left second molar (tooth 75),The buccal surface of the mandibular left central incisor (tooth 71),The lingual surface of the mandibular right second molar (tooth 85). Each surface will take a score from 0-3. The scores of the involved surfaces will be totaled and divided by the number of teeth scored to get the index value.
Oral hygiene index (OHI-S) assessment | 6 weeks
  For primary dentition, the modified version of the OHI-S by Miglani et al will be used, it is divided into two scores debris index and calculus index only the debris index will be used in which the index teeth are: The buccal surface of maxillary right second molar (tooth 55), The buccal surface of the maxillary right central incisor (tooth 51), The buccal surface maxillary left second molar (tooth 65), The lingual surface of the mandibular left second molar (tooth 75),The buccal surface of the mandibular left central incisor (tooth 71),The lingual surface of the mandibular right second molar (tooth 85). Each surface will take a score from 0-3. The scores of the involved surfaces will be totaled and divided by the number of teeth scored to get the index value.
Oral hygiene index (OHI-S) assessment | 18 weeks
  For primary dentition, the modified version of the OHI-S by Miglani et al will be used, it is divided into two scores debris index and calculus index only the debris index will be used in which the index teeth are: The buccal surface of maxillary right second molar (tooth 55), The buccal surface of the maxillary right central incisor (tooth 51), The buccal surface maxillary left second molar (tooth 65), The lingual surface of the mandibular left second molar (tooth 75),The buccal surface of the mandibular left central incisor (tooth 71),The lingual surface of the mandibular right second molar (tooth 85). Each surface will take a score from 0-3. The scores of the involved surfaces will be totaled and divided by the number of teeth scored to get the index value.
Oral hygiene index (OHI-S) assessment | 30 weeks
  For primary dentition, the modified version of the OHI-S by Miglani et al will be used, it is divided into two scores debris index and calculus index only the debris index will be used in which the index teeth are: The buccal surface of maxillary right second molar (tooth 55), The buccal surface of the maxillary right central incisor (tooth 51), The buccal surface maxillary left second molar (tooth 65), The lingual surface of the mandibular left second molar (tooth 75),The buccal surface of the mandibular left central incisor (tooth 71),The lingual surface of the mandibular right second molar (tooth 85). Each surface will take a score from 0-3. The scores of the involved surfaces will be totaled and divided by the number of teeth scored to get the index value.
Visio-tactile evaluation of the white spot lesion | Baseline
  Using a dental light reflector, visual inspection of all tooth surfaces for WSLs will be undertaken, with wet tooth surfaces and again after 5 seconds of drying with a gentle air stream. Each lesion will be scored according to ICDAS II criteria for severity, selecting only lesions scored as 1, 2 or 3.
Visio-tactile evaluation of the white spot lesion | 6 weeks
  Using a dental light reflector, visual inspection of all tooth surfaces for WSLs will be undertaken, with wet tooth surfaces and again after 5 seconds of drying with a gentle air stream. Each lesion will be scored according to ICDAS II criteria for severity, selecting only lesions scored as 1, 2 or 3.
Visio-tactile evaluation of the white spot lesion | 18 weeks
  Using a dental light reflector, visual inspection of all tooth surfaces for WSLs will be undertaken, with wet tooth surfaces and again after 5 seconds of drying with a gentle air stream. Each lesion will be scored according to ICDAS II criteria for severity, selecting only lesions scored as 1, 2 or 3.
Visio-tactile evaluation of the white spot lesion | 30 weeks
  Using a dental light reflector, visual inspection of all tooth surfaces for WSLs will be undertaken, with wet tooth surfaces and again after 5 seconds of drying with a gentle air stream. Each lesion will be scored according to ICDAS II criteria for severity, selecting only lesions scored as 1, 2 or 3.
White spot lesion evaluation using DIAGNOdent | Baseline
  Probe B OF Laser fluorescence (LF) examination for each lesion will be performed using DIAGNOdent. It operates with a diode laser having a wavelength of 655 nm and 1 mW peak power. Sound enamel does not fluoresce at this wavelength, but caries and bacteria do. The instrument is calibrated according to manufacturer's instructions. A baseline zero value for each patient is obtained by choosing a clear non carious patch of enamel usually middle third of an anterior tooth. By pointing the pen perpendicular to this area and touching the set button for 2 seconds until set 0 appears, the button is then released. Zero baseline value has been set. Under cotton roll isolation and after air drying with an air syringe, the DIAGNOdent probe will be placed perpendicular to the test site and rotated along the lesion to scan the area completely. Three measurements of each lesion will be taken and averaged to give the final score.
White spot lesion evaluation using DIAGNOdent | 6 weeks
  Probe B OF Laser fluorescence (LF) examination for each lesion will be performed using DIAGNOdent. It operates with a diode laser having a wavelength of 655 nm and 1 mW peak power. Sound enamel does not fluoresce at this wavelength, but caries and bacteria do. The instrument is calibrated according to manufacturer's instructions. A baseline zero value for each patient is obtained by choosing a clear non carious patch of enamel usually middle third of an anterior tooth. By pointing the pen perpendicular to this area and touching the set button for 2 seconds until set 0 appears, the button is then released. Zero baseline value has been set. Under cotton roll isolation and after air drying with an air syringe, the DIAGNOdent probe will be placed perpendicular to the test site and rotated along the lesion to scan the area completely. Three measurements of each lesion will be taken and averaged to give the final score.
White spot lesion evaluation using DIAGNOdent | 18 weeks
  Probe B OF Laser fluorescence (LF) examination for each lesion will be performed using DIAGNOdent. It operates with a diode laser having a wavelength of 655 nm and 1 mW peak power. Sound enamel does not fluoresce at this wavelength, but caries and bacteria do. The instrument is calibrated according to manufacturer's instructions. A baseline zero value for each patient is obtained by choosing a clear non carious patch of enamel usually middle third of an anterior tooth. By pointing the pen perpendicular to this area and touching the set button for 2 seconds until set 0 appears, the button is then released. Zero baseline value has been set. Under cotton roll isolation and after air drying with an air syringe, the DIAGNOdent probe will be placed perpendicular to the test site and rotated along the lesion to scan the area completely. Three measurements of each lesion will be taken and averaged to give the final score.
White spot lesion evaluation using DIAGNOdent | 30 weeks
  Probe B OF Laser fluorescence (LF) examination for each lesion will be performed using DIAGNOdent. It operates with a diode laser having a wavelength of 655 nm and 1 mW peak power. Sound enamel does not fluoresce at this wavelength, but caries and bacteria do. The instrument is calibrated according to manufacturer's instructions. A baseline zero value for each patient is obtained by choosing a clear non carious patch of enamel usually middle third of an anterior tooth. By pointing the pen perpendicular to this area and touching the set button for 2 seconds until set 0 appears, the button is then released. Zero baseline value has been set. Under cotton roll isolation and after air drying with an air syringe, the DIAGNOdent probe will be placed perpendicular to the test site and rotated along the lesion to scan the area completely. Three measurements of each lesion will be taken and averaged to give the final score.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed I Mekky, BDS, Principal Investigator — Alexandria University; Karin ML Dowidar, PhD, Study Director — Alexandria University; Dalia AM Talaat, PhD, Study Director — Alexandria University
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Egypt

REFERENCES:
- [Background] Willmot DR. White lesions after orthodontic treatment: does low fluoride make a difference? J Orthod. 2004 Sep;31(3):235-42; discussion 202. doi: 10.1179/146531204225022443. PMID 15489367
- [Background] Llena C, Leyda AM, Forner L. CPP-ACP and CPP-ACFP versus fluoride varnish in remineralisation of early caries lesions. A prospective study. Eur J Paediatr Dent. 2015 Sep;16(3):181-6. PMID 26418918
- [Background] Cochrane NJ, Shen P, Yuan Y, Reynolds EC. Ion release from calcium and fluoride containing dental varnishes. Aust Dent J. 2014 Mar;59(1):100-5. doi: 10.1111/adj.12144. Epub 2014 Feb 4. PMID 24494654
- [Background] Ismail AI, Sohn W, Tellez M, Amaya A, Sen A, Hasson H, Pitts NB. The International Caries Detection and Assessment System (ICDAS): an integrated system for measuring dental caries. Community Dent Oral Epidemiol. 2007 Jun;35(3):170-8. doi: 10.1111/j.1600-0528.2007.00347.x. PMID 17518963
- [Background] Miglani DC, Beal JF, James PM, Behari SA. The assessment of dental cleanliness status of the primary dentition using a modification of the simplified oral hygiene index(OHIS-M). J Indian Dent Assoc. 1973 Dec;45(12):385-8. No abstract available. PMID 4535076
- [Background] Braga MM, Mendes FM, Ekstrand KR. Detection activity assessment and diagnosis of dental caries lesions. Dent Clin North Am. 2010 Jul;54(3):479-93. doi: 10.1016/j.cden.2010.03.006. PMID 20630191